CLINICAL TRIAL: NCT02200276
Title: Influenza Immunization in Adults Over Age 75
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NA_00092365
Record Dates: First submitted 2014-07-11; First posted 2014-07-25 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Influenza; Immunization; Older Adults; Over Age 75
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Influenza Immunization (Other): Influenza immunization in adults over age 75
  Interventions: Biological: Influenza

INTERVENTIONS:
Biological: Influenza

SUMMARY:
The immune system is the part of the body that protects against infection. The immune system often doesn't work as effectively as people get older. This research is being done to find out how the immune systems in older people who are over age 75 respond to influenza vaccine (flu shot). We also want to find out if chronic cytomegalovirus (CMV) infection, a common virus infection in older persons affects the immune response in people older than 75 years of age who receive a flu shot. The Flu Shot is a vaccine approved for the prevention of influenza ("Flu") infections and is recommended every year for all persons 50 years and older. People who are older than 75 years of age are considered healthy or frail may join. A total of 1025 persons will be participating in this study.

In order to determine if you are qualified for the study, we would ask you to answer a few questions over the phone that will take approximately 5 minutes. If you qualify and agree to proceed, you will be asked to come to Johns Hopkins Bayview Medical Center or, if you are unable to come to Bayview, one of our staff can visit you at your home. During that visit we obtain consent, review your medical history, and measure your vital signs, walking speed and grip strength. We will also administer a few brief questionnaires and collect urine and blood samples. We will then give you the Influenza vaccine for free. 7 days post receiving your Influenza Vaccine we will collect a small blood sample for further immune system testing. also, you will be asked to complete a 12-question survey which will assess your symptoms over the past 7 days (post receiving the Influenza vaccine). Also 4 weeks post receiving your Influenza vaccine you will be asked to complete a third visit that will include follow up health questionnaires and an influenza symptoms assessment questionnaire and vital signs. A third blood draw will be collected (approximately 10 teaspoons) to measure immune responses to the influenza vaccine. In addition, you will receive your test result (CBC/w/Diff.) from visit #1. Throughout the influenza study season, we will call you once a week to ask about your general health and any Flu-like symptoms. These calls will be made throughout the Flu season which typically lasts through May. If you begin to have any influenza like symptoms at any time during the study, we ask that you call our office to report these symptoms so that we may perform vital signs, nasal swab to confirm influenza, and a fourth blood draw to look at the immune response and protection of influenza vaccine.

DETAILED DESCRIPTION:
Seasonal influenza causes significant morbidity and mortality and is the fourth leading cause of death for older Americans. Annual immunization with a trivalent inactivated influenza vaccine (TIV) is recommended for all adults 50 years and older. However, despite improved vaccination coverage in older adults over time, influenza-related mortality has actually increased. While many TIV studies indicate its benefit for older adults as a whole, these studies lacked representation of the older and frail subset of the elderly who suffer over three-quarters of influenza-related mortality. Our pilot study funded by a Beeson K23 award showed significant vaccine failures in both antibody response to TIV and clinical protection in the frail elderly. Our preliminary data also suggest that chronic cytomegalovirus (CMV) infection as defined by the presence of CMV viral DNA in peripheral monocytes using a highly sensitive and specific nested PCR-based assay developed in our laboratory, rather than anti-CMV IgG serology, is associated with poor antibody and T-cell responses to TIV immunization as well as poor clinical protection. This is likely because anti-CMV IgG serology, the conventional diagnostic measure for chronic CMV infection, is a crude measure that merely indicates prior exposure to CMV and does not distinguish chronic (persistent) from past (resolved) infections. Mechanistically, precipitous immune functional decline has been observed in those over 75 and chronic CMV infection may contribute significantly to age-related immune senescent remodeling, termed immunosenescence. In order to improve our assessment of the effectiveness of TIV immunization and understanding of risk factors and underlying immune mechanisms that determine vaccine failure in adults over age 75, the frail, oldest old adult subset, this study is designed to conduct prospective, 4-year TIV immunization and post-vaccination influenza surveillance in adults over 75 years. We will first assess chronic CMV infection defined by detectable CMV DNA in peripheral blood monocytes and frailty status of the study participants and administer the Fluzone High-Dose TIV vaccine. Influenza-like illness (ILI) cases will be identified through post-vaccination influenza surveillance as previously done in the Beeson project and respiratory specimens obtained from ILI cases will be tested using the cutting edge PCR-based IBIS assay which can accurately subtype influenza and other respiratory viruses in the laboratory of Dr. Charlotte Gaydos in Division of Infectious Disease, a co-investigator of this project. Strain-specific antibody responses to TIV immunization will be measured by the standard hemogglutination inhibition (HI) assay. We will also evaluate T-cell responses to influenza viruses at baseline and after TIV immunization. Taken together, these studies will provide more accurate assessment of the clinical effectiveness of TIV immunization in real world geriatric population over age 75 and its underlying humoral and cell-mediated immune mechanisms. Moreover, we investigate the role of chronic CMV infection as defined by the presence of CMV viral DNA in peripheral monocytes as a risk factor for vaccine failure in the elderly over age 75. Because this oldest old subset is growing most rapidly in numbers and is at greatest risk for influenza-related morbidity and mortality. The long-term goal of this research is to strengthen immune protection against influenza for vulnerable older Americans through more effective and targeted immunization strategies as well as possibly through prevention and mitigation of chronic CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 75 years

Exclusion Criteria:

* Allergies to egg or vaccine
* Active malignancies
* On radiation or chemotherapy
* Active systemic inflammatory diseases including rheumatoid arthritis, Crohn's disease, and ulcerative colitis
* Acute exacerbation of chronic cardiopulmonary conditions including decompensated CHF or COPD
* Taking oral steroids (such as prednisone) or immune modulating drugs (such as methotrexate).
* Lacking the capacity to consent (individuals who do not understand what Flu shot is or need someone else to decide if s/he should get the Flu shot)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1025 (Estimated)
Dates: Start 2014-03; Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Presence of CMV Viral DNA in Peripheral Blood Monocytes | At the end of each flu season for the next 4 years
  To assess the role of chronic CMV infection as defined by presence of CMV viral DNA in peripheral monocytes as a risk factor for vaccine failure in this oldest old subset.

SECONDARY OUTCOMES:
Immune Responses to High Dose TIV Immunization | At the end of the study-5th year

OTHER OUTCOMES:
Effectiveness of High Dose TIV Immunization | At the end of the study, 5th year
  To assess clinical effectiveness of High Dose TIV immunization in real world geriatric population over age 75 through post-vaccination influenza detection
Influence of Frailty and Chronic CMV Infection on Vaccine-Induced Influenza Strain-Specific Antibody Titers and T-Cell Responses | At the end of the study, 5th year
  To assess potential interaction between chronic CMV infection as defined above and frailty in their impact on antibody and T-cell responses to as well as clinical protection of High Dose TIV immunization in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Leng, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University; JHAAC 5501 Hopkins Bayview Circle, 1B84, Baltimore, Maryland, United States